CLINICAL TRIAL: NCT06804980
Title: The DEterminig Statin Intolerance for Rosuvastatin Trial
Brief Title: DESIFOR-EXPAND (MHIF)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2236054
Record Dates: First submitted 2025-01-23; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Statin Therapy; Statin Adverse Reaction; Statin
Keywords: Statin Intolerance; lipid-lowering medication; LDL; LDL Cholesterol
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Each kit will include 3 28-day packs of placebo and 2 28-day packs of rosuvastatin, assigned at random. Each kit will have a unique identification number, which the pharmacy will record in a drug tracking log as it is dispensed. Within each kit, a unique identifying number will be present on each blister pack which can be used to determine the order of allocation of placebo and rosuvastatin.
Who Masked: Participant, Care Provider, Investigator
Masking Description: There will be unblinded and blinded research staff. Unblinding for the patient and provider will occur at 6-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo taken first, drug taken second (Other): The placebo is assigned to the patient first, with the medication taken in the second part of participation.
  Interventions: Drug: Rosuvastatin (Crestor); Drug: Placebo
- Drug taken first, then placebo taken second (Other): The placebo is assigned to the patient first, with the medication taken in the second part of participation.
  Interventions: Drug: Rosuvastatin (Crestor); Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin (Crestor) — The patient will take 3 28-day packs of placebo and 2 28-day packs of rosuvastatin. The order in which they take the placebo or rosuvastatin will be assigned at random.
Drug: Placebo — The patient will take 3 28-day packs of placebo and 2 28-day packs of rosuvastatin. The order in which they take the placebo or rosuvastatin will be assigned at random.

SUMMARY:
The DESIFOR pilot study was conducted to determine the feasibility of utilizing an n-of-1 trial to facilitate tolerance of unblinded rosuvastatin in patients with prior statin intolerance

DETAILED DESCRIPTION:
Recently developed lipid lowering therapies have been shown to significantly reduce LDL cholesterol and subsequent CVD risk (1, 2). However, they are expensive, and the cost-effectiveness of these medications remains controversial, especially in primary prevention. Novel lipid lowering therapies are frequently considered for individuals with statin intolerance, but payers frequently deny prescription for these medications due to lack of adequate proof of true statin intolerance. How to accurately determine statin intolerance remains a clinical conundrum for both patients and providers. A more scientific, definitive method to determine statin intolerance could potentially allow appropriate, cost-effective use of statin therapy in individuals found to not actually be statin intolerant as well as judicious use of novel medications in patients who are found to truly be statin intolerant.

The DESIFOR pilot study was conducted to determine the feasibility of utilizing an n-of-1 trial to facilitate tolerance of unblinded rosuvastatin in patients with prior statin intolerance. The DESIFOR pilot study was a single-center, randomized, double-blinded, n-of-1 trial in patients aged 21 to 79 years and eligible for statin therapy by current guidelines but not on therapy due to intolerance of >2 statins. Using a double-blinded, N-of-1 randomized trial in patients with previous statin intolerance, <10% of patients had data suggestive of true statin intolerance, and 2/3 of patients were subsequently able to tolerate 3-months of unblinded treatment with rosuvastatin (3). These data raise the hypothesis that an n-of-1 trial can be used to facilitate tolerance of unblinded rosuvastatin in patients with prior statin intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 21 years old) with a prior history of statin intolerance. Statin intolerance is defined by discontinuation of at least 2 different statin medications due to possible side effects. Patients can participate in the trial while on other lipid-lowering agents, such as ezetimibe and PSCK9 inhibitors, as long as the patient has been on the other lipid lowering therapy and tolerating it well for at least 1 month. For individuals with established ASCVD or multiple ASCVD risk factors, initiation of other lipid lowering therapy prior to participation in DESIFOR is encouraged.
* 2. At least 30 days since discontinued use of a statin

Exclusion Criteria:

* Women who are pregnant, nursing or attempting to become pregnant
* Individuals who experienced severe reactions in the past, including rhabdomyolysis, severe myositis, anaphylaxis
* Individuals who are not otherwise clinically indicated to take rosuvastatin 20 mg

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal symptom presence/absence | 9 months
  To determine the prevalence of true statin intolerance, defined by a statistical difference in the mean musculoskeletal symptom score while on statin therapy compared to placebo, in patients previously identified as statin intolerant.
Statin Tolerance | 9 months
  To determine the prevalence of statin tolerance, defined as continuous use of 3 months of unblinded rosuvastatin, in individuals with previous statin intolerance but without evidence of true statin intolerance in the DESIFOR protocol.
Variables associated with statin intolerance | 9 months
  To determine the clinical variables associated with true statin intolerance.

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis Heart Institute Foundation, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No